CLINICAL TRIAL: NCT03037541
Title: A Single-Center, Randomized, Single-Blinded, Placebo-Controlled Trial on the Efficacy of Cryosurgery and 5-Fluorouracil 0.5% Cream Combination Therapy for the Treatment of Actinic Keratosis
Brief Title: Cryosurgery and Cream Combination for Actinic Keratosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00014209
Record Dates: First submitted 2011-09-08; First posted 2017-01-31 (Estimated); Results first posted 2017-03-23 (Actual); Last update posted 2018-08-29 (Actual); Status verified 2018-07

CONDITIONS: Actinic Keratosis
Keywords: Wake Forest; Actinic Keratosis; Cryosurgery; Cream
MeSH Terms: conditions — Keratosis, Actinic | interventions — cetyl alcohol, propylene glycol, sodium lauryl sulfate non-lipid cleansing lotion

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1 Carac (fluorouracil) 0.5% cream (Experimental): Carac cream (fluorouracil) 0.5% applied daily on the face for one week
  Interventions: Drug: Carac Cream
- Group 2 Placebo (Placebo Comparator): Placebo Cetaphil cream applied daily on the face for one week
  Interventions: Drug: Placebo Cetaphil cream

INTERVENTIONS:
Drug: Carac Cream — Carac Cream will be used once daily for seven consecutive days
  Arms: Group 1 Carac (fluorouracil) 0.5% cream
Drug: Placebo Cetaphil cream — Placebo Cetaphil Cream will be used once daily for seven consecutive days
  Other Names: Cetaphil
  Arms: Group 2 Placebo

SUMMARY:
Carac 0.5% cream is approved for daily topical treatment of AK's for up to four weeks as tolerated, though local irritation often occurs within the first week of treatment and increases in a dose-dependent manner. In this study, the investigators will examine the combination of standard cryosurgery treatment followed by a shortened course of topical fluorouracil cram. The investigators anticipate that a one week treatment course will maintain overall effectiveness when combined with previous cryosurgery, but will reduce the overall adverse effects of topical therapy due to the reduced treatment time and the presence of fewer baseline lesions to treat. This treatment approach may provide a more acceptable risk/benefit ratio option for patients with more extensive disease and simplify standard combination treatment options. The primary objective is to evaluate the efficacy of combination cryosurgery and 5-fluorouracil0.5% cream, compared to combination cryosurgery and placebo in the treatment of actinic keratosis lesions. The efficacy of this combination therapy will be evaluated by assessing AK lesion clearance. The primary efficacy parameter will be 10% clearance of all AK lesions from treatment initiation to end-of-treatment.

DETAILED DESCRIPTION:
This is a randomized (1:1), single-blind, placebo controlled, single center prospective study. Subjects will first undergo cryosurgery of all clinically apparent AK lesions, limited to the face or balding scalp. Three weeks after cryosurgery, subjects will then be randomized (1:1 according to standard randomization tables) and directed to apply either Carac 0.5% cream or placebo cream (Cetaphil Cream) to the face or balding scalp at bedtime for seven consecutive days, washed off each following morning. Each does of study cream will be applied at approximately the same time of day and will remain on the skin for approximately eight hours. Subject evaluation, Investigator Global Assessments, Quality of Life lesion counts and photography shall be performed at Baseline. At Week 3, study drug will be dispensed and the global assessments and assessment of improvement will be performed. A Medication Tolerability Assessment will occur at Week 4 when the study drug will be returned. Investigator Global Assessment, lesion count, Global Assessment of Improvement and Quality of Life will be measured at Week 8 and Week 26 (or end of study). Photography will be done at Week 26 or end of study.

ELIGIBILITY:
Inclusion Criteria:

* Must be male or female and at least 18 years of age. Each subject must demonstrate good health as determined by a baseline medical history.
* Female subjects myst be of either non-childbearing potential, or childbearing potential provided: negative urine pregnancy test and using two acceptable methods of effective contraception (abstinence, birth control pills.patch, DepoProvera, tubal ligation, vasectomy of the partner in a monogamous relationship, condoms and spermicidal form or gel and/or cervical cap or sponge), as determined by the investigator
* At least eight clinically typical, visible and discrete AK lesions within the treatment area on the face or balding scalp
* Subjects must be able and willing to comply with study procedures and have provided written informed consent.

Exclusion Criteria:

* Cosmetic or therapeutic procedures (e.g., use of liquid nitrogen, surgical excision, curettage, dermabrasion, medium or greater depth chemical peel, laser resurfacing) within the selected treatment area in the previous four weeks.
* Treatment with systemic medications that suppress the immune system within the previous four weeks.
* Field treatments with topical 5-FU, imiquimod, diclofenac, or photodynamic therapy, or more widespread field treatment with dermabrasion, medium or greater depth chemical peel, or laser resurfacing within the previous six months.
* Any known dihydropyrimidine dehydrogenase enzyme deficiency.
* In addition, subjects who have any skin condition or disease that may require concurrent therapy or may confound the evaluation as determined by the investigator, or a history of hypersensitivity to any of the formulation components will be excluded from study.
* Subjects may not use other topical agents such as glycolic acid products, alpha-hydroxy acid products, retinoids and chemical peel agents on teh treatment area while on study. The use of these products are not allowed four weeks prior to study enrollment. Introduction of any other prescription medication, topical or systemic for actinic keratosis while participating in the study is not permitted.
* Pregnant women, women who are breast feeding, or women of childbearing potential who are not practicing two acceptable methods of effective contraception.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-01-05 (Actual); Primary Completion 2013-10-29 (Actual); Study Completion 2013-10-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Jorizzo, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences Department of Dermatology, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 1 Carac (Fluorouracil) 0.5% Cream | Group 2 Placebo
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 Carac (Fluorouracil) 0.5% Cream | Group 2 Placebo | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 8 | 17
  >=65 years | 21 | 22 | 43
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 27 | 28 | 55
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 30 | 29 | 59
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 30 | 30 | 60
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Number Participants With 100% Clearance
Description: The primary endpoint is number of participants that receive 100% clearance of AK lesions from treatment initiation to end of treatment
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 Carac (Fluorouracil) 0.5% Cream | Group 2 Placebo
Number analyzed (Participants) | 30 | 30
Participants | 12 | 13

2. Secondary Outcome: Number of Participants With 75% Clearance
Description: The secondary endpoint is number of participants that receive 75 % clearance of
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 Carac (Fluorouracil) 0.5% Cream | Group 2 Placebo
Number analyzed (Participants) | 30 | 30
Participants | 18 | 16

ADVERSE EVENTS:
Arm/Group | Group 1 Carac (Fluorouracil) 0.5% Cream | Group 2 Placebo
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 4/30 | 5/30
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 Carac (Fluorouracil) 0.5% Cream (N=30) | Group 2 Placebo (N=30)
basal cell carcinoma (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
joint pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
viral infection (Infections and infestations) | 0 (0) | 3 (3)
tooth pain (Infections and infestations) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes